CLINICAL TRIAL: NCT07175766
Title: A Study on the Lipid-Modulating and Health Benefits of Dachundou No Sugar Added Soymilk in Humans
Brief Title: Dachundou No Sugar Added Soymilk for Lipid Modulation
Acronym: DNS Soymilk
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Responsible Party: Principal Investigator, Chi-Chang Huang, Distinguished Professor, National Taiwan Sport University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-25-058-A2; 2025-Dachundou-IRB-25-058-A2 (Other: WEI CHUAN FOODS CORPORATION)
Record Dates: First submitted 2025-09-02; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Dyslipidemias; Hypercholesterolemia; Cardiovascular Diseases
Keywords: Soy milk; Dachundou; No sugar added soymilk; Cholesterol; Total cholesterol; LDL cholesterol; HDL cholesterol; Lipid metabolism; Functional food; Cardiovascular health
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: This is a single-group, open-label interventional study. All participants meeting the eligibility criteria will receive the same intervention: daily supplementation with Dachundou No Sugar Added Soymilk (2 bottles of 375 mL each; total 750 mL/day) for 8 consecutive weeks. No control or placebo group will be included. Outcomes will be assessed at baseline (week -2 and week 0), mid-intervention (week 4), end of intervention (week 8), and follow-up (week 10).
Masking Description: This study is conducted as an open-label, single-group dietary intervention. No masking is applied to participants, investigators, care providers, or outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Soymilk Intervention (Experimental): Participants will consume two bottles of Dachundou No Sugar Added Soymilk daily (375 mL each; total 750 mL per day) for 8 consecutive weeks. Assessments will be performed at baseline (week -2 and week 0), during the intervention (week 4 and week 8), and post-intervention (week 10).
  Interventions: Dietary Supplement: Dachundou No Sugar Added Soymilk

INTERVENTIONS:
Dietary Supplement: Dachundou No Sugar Added Soymilk — Participants will consume two bottles of Dachundou No Sugar Added Soymilk daily (375 mL each; total 750 mL per day) for 8 consecutive weeks. The product is packaged in 375 mL cartons and made from non-GMO soybeans, containing approximately 4.2 g of soy protein per 100 mL. The soymilk is unsweetened and stored at 0-7°C.
  Other Names: Unsweetened Dachundou Soymilk

SUMMARY:
Cardiovascular disease is one of the leading causes of death worldwide, and high cholesterol is a major risk factor. Diet is known to play an important role in managing blood lipids. Soy milk is a common plant-based drink rich in protein and isoflavones, which may help lower cholesterol and improve heart health.

This clinical trial will evaluate whether daily consumption of Dachundou No Sugar Added Soymilk can help reduce cholesterol levels in adults with elevated total cholesterol (≥200 mg/dL). A total of 50 participants aged 18-65 will be recruited. Participants will drink two bottles of soymilk per day (375 mL each, total 750 mL) for 8 weeks.

During the study, researchers will measure cholesterol, blood pressure, body weight, waist circumference, and other health indicators. The results will help determine whether Dachundou No Sugar Added Soymilk can improve blood lipid levels and contribute to cardiovascular health.

DETAILED DESCRIPTION:
Cardiovascular disease remains a leading cause of morbidity and mortality worldwide, with dyslipidemia being one of the most important risk factors. Dietary interventions, such as plant-based proteins and bioactive compounds, have been shown to improve lipid profiles and reduce cardiovascular risk. Soy milk is widely consumed in Asia and contains soy protein and isoflavones, which have antioxidant, anti-inflammatory, and lipid-regulating effects.

Previous studies suggest that soy protein may lower total cholesterol and LDL-C through inhibition of HMG-CoA reductase and upregulation of LDL receptor expression, while soy isoflavones may enhance lipid metabolism and endothelial function through estrogen-like actions.

This trial aims to evaluate the lipid-lowering efficacy of Dachundou No Sugar Added Soymilk in adults with fasting total cholesterol ≥200 mg/dL. A total of 50 participants, aged 18-65 years, non-smokers, without alcohol abuse, and otherwise healthy, will be enrolled. All participants will consume two bottles of soymilk per day (375 mL each; total 750 mL) for 8 consecutive weeks.

Assessments will be performed at baseline (week -2 and week 0), during the intervention (week 4 and week 8), and post-intervention (week 10). Measurements include anthropometrics (height, weight, waist circumference, blood pressure), blood biochemistry (lipid profile, glucose, liver and kidney function), oxidative stress (oxidized LDL via TBARS), and lifestyle factors (dietary records and physical activity questionnaires).

The primary outcome is the change in total cholesterol from baseline to week 8. Secondary outcomes include changes in LDL-C, HDL-C, triglycerides, oxidized LDL, liver/kidney function, and anthropometric indices. The findings will provide evidence on whether Dachundou No Sugar Added Soymilk can serve as a dietary intervention to improve blood lipid levels and promote cardiovascular health.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* Fasting total cholesterol (TC) ≥200 mg/dL at both screening (week -2) and baseline (week 0)
* Non-smokers
* No alcohol abuse
* Able and willing to comply with study procedures, dietary restrictions, and follow-up visits

Exclusion Criteria:

* Pregnant or lactating women
* Menopausal or postmenopausal women
* Diagnosed with chronic diseases under medical treatment (e.g., hypertension, hyperlipidemia, diabetes, liver, kidney, gastrointestinal, cardiovascular disease, cancer)
* Use of dietary supplements or drugs affecting lipid metabolism within 1 month before study entry or during the study
* Cognitive impairment preventing informed consent or protocol compliance
* History of allergy to soy milk, oats, or gluten-containing products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in total cholesterol (TC) | Baseline (week 0) to week 8
  Serum total cholesterol concentration will be measured using an automated biochemical analyzer to evaluate the lipid-lowering efficacy of Dachundou No Sugar Added Soymilk.

SECONDARY OUTCOMES:
Change in LDL cholesterol (LDL-C) | Baseline to week 8
  LDL-C concentration measured by automated biochemical analyzer.
Change in HDL cholesterol (HDL-C) | Baseline to week 8
  HDL-C concentration measured by automated biochemical analyzer.
Change in triglycerides (TG) | Baseline to week 8
  Serum triglyceride concentration measured by automated biochemical analyzer.
Change in oxidized LDL (TBARS assay) | Baseline to week 8
  Oxidative stress marker (TBARS values in LDL fraction).
Change in body weight (kg) | Baseline, week 4, week 8, week 10
  Weight will be measured using a calibrated digital scale, with participants wearing light clothing and no shoes.
Liver function markers (AST, ALT, γ-GT) | Baseline and week 8
  Serum liver enzymes assessed for safety.
Kidney function markers (BUN, creatinine, uric acid) | Baseline and week 8
  Serum renal parameters assessed for safety.
Change in dietary intake (kcal/day) | Baseline, week 4, week 8, week 10
  Dietary intake will be assessed using 3-day food records analyzed with nutrition analysis software to calculate average daily energy intake (kcal/day).
Change in body mass index (BMI, kg/m²) | Baseline, week 4, week 8, week 10
  BMI will be calculated as weight in kilograms divided by height in meters squared.
Change in waist circumference (cm) | Baseline, week 4, week 8, week 10
  Waist circumference will be measured at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest, using a standard tape measure.
Change in blood pressure (mmHg) | Baseline, week 4, week 8, week 10
  Systolic and diastolic blood pressure will be measured using an automated sphygmomanometer after 5 minutes seated rest.
Change in physical activity level (IPAQ-SF score, MET-min/week) | Baseline, week 4, week 8, week 10
  Physical activity will be assessed using the International Physical Activity Questionnaire - Short Form (IPAQ-SF). Scores will be calculated as MET-minutes per week. Higher scores indicate greater physical activity levels.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Sport University, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the trial involves sensitive health-related data collected from human participants. Only aggregated and de-identified summary results will be published in scientific journals and conference presentations.

REFERENCES:
- [Background] Ramdath DD, Padhi EM, Sarfaraz S, Renwick S, Duncan AM. Beyond the Cholesterol-Lowering Effect of Soy Protein: A Review of the Effects of Dietary Soy and Its Constituents on Risk Factors for Cardiovascular Disease. Nutrients. 2017 Mar 24;9(4):324. doi: 10.3390/nu9040324. PMID 28338639